CLINICAL TRIAL: NCT03974984
Title: Anesthesia and Immunological and Oxidative Stress in Relation to Abdominal Cancer Surgery
Acronym: ANIMOX
Status: Withdrawn | Type: Observational
Why Stopped: Not feasable due to logistics
Sponsor: University of Copenhagen (Other)
Responsible Party: Principal Investigator, Rune Børch Hasselager, Medical Doctor, University of Copenhagen
Other Study IDs: SJ-704
Record Dates: First submitted 2019-05-31; First posted 2019-06-05 (Actual); Last update posted 2020-11-05 (Actual); Status verified 2020-11

CONDITIONS: Anesthesia; Colon Cancer; Surgery
MeSH Terms: conditions — Colonic Neoplasms | interventions — Anesthesia, Epidural; Anti-Inflammatory Agents, Non-Steroidal

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Standard blood samples analyzed immediately after sampling. These include Hgb, Leucocytes including a differential count, thrombocytes, ALAT, LDH, Alkaline phosphatase, bilirubin, INR, albumin, Na, K, Creatinine, CRP and Glucose.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- The "Hvidovre population":: We will include patients undergoing laparoscopic hemicolectomy for cancer scheduled for anesthesia with total intravenous anesthesia combined with epidural anesthesia and perioperative NSAID on Hvidovre Hospital.
  Interventions: Procedure: Colon Resection; Procedure: Epidural anesthesia; Drug: NSAID
- The "Zealand University Hospital population": The immunological and oxidative stress in relation to abdominal surgery (IMOX) study is ongoing at Zealand University Hospital, Roskilde. It is a prospective explorative study cohort that consists of 60 patients undergoing laparoscopic colorectal cancer surgery.
  The population has been anesthetized according to the standard operating procedure with either total intravenous anesthesia with propofol and remifentanil or volatile anesthesia with sevoflurane combined with a fast acting opioid (remifentanil or sufentanil). Patients anaesthetized with other techniques including epidural or other regional blocks will be excluded from the analysis.
  Interventions: Procedure: Colon Resection

INTERVENTIONS:
Procedure: Colon Resection — All patients undergo laparoscopic colon cancer resection.
Procedure: Epidural anesthesia — Epidural inserted preoperatively and kept for 1 day postoperatively
  Groups: The "Hvidovre population":
Drug: NSAID — NSAID administered according to standard operating procedure postoperatively
  Groups: The "Hvidovre population":

SUMMARY:
Colorectal cancer is a frequent type of cancer accounting for 600,000 deaths annually. Surgical resection remains the best treatment for long-term survival. However, studies suggest that events in the perioperative period can induce metastasis formation and tumor growth. Tumor cells are released into the blood stream during surgery and the surgical stress may create a favorable environment for dissemination of tumor cells into distant tissue. This is done by a cascade of pro-cancerous catecholamines, prostaglandins and cytokines combined with an impaired anti-cancerous cell mediated immune response.

Until recently, focus on the anesthetic management of cancer patients has been limited. Relatively small alterations in the perioperative anesthetic management may play a tremendous role in tumor progression. Optimizing anesthesia to reduce the surgical stress response could improve recurrence rates and long-term outcomes for cancer patients by inhibiting perioperative metastasis formation. Regional anesthesia and amide local anesthetics are suspected to calm the immunologic storm of prostaglandins, catecholamines and cytokines when used in the perioperative phase. Furthermore, volatile inhalational anesthesia is thought to modulate the immune system in a pro-cancerous way, while propofol may have opposite effects. Many of these recent studies are statistically underpowered and susceptible to bias, and experts in cancer treatment and anesthesia have emphasized the need for further research within this specific field.

In this study the investigators aim to characterize differences in the immunologic response to surgery between inhalational, total intravenous and epidural anesthesia. This will be done by analyzing blood samples obtained in the perioperative period in patients undergoing different modes of anesthesia. The Investigators will furthermore describe the quality of recovery for patients anesthetized with the different methods

DETAILED DESCRIPTION:
Background and Purpose Colorectal cancer is a frequent type of cancer accounting for 600,000 deaths annually. Surgical resection remains the best treatment for long-term survival. However, studies suggest that events in the perioperative period can induce metastasis formation and tumor growth. Tumor cells are released into the blood stream during surgery and the surgical stress may create a favorable environment for dissemination of tumor cells into distant tissue. This is done by a cascade of pro-cancerous catecholamines, prostaglandins and cytokines combined with an impaired anti-cancerous cell mediated immune response.

Until recently, focus on the anesthetic management of cancer patients has been limited. Relatively small alterations in the perioperative anesthetic management may play a tremendous role in tumor progression. Optimizing anesthesia to reduce the surgical stress response could improve recurrence rates and long-term outcomes for cancer patients by inhibiting perioperative metastasis formation. Regional anesthesia and amide local anesthetics are suspected to calm the immunologic storm of prostaglandins, catecholamines and cytokines when used in the perioperative phase. Furthermore, volatile inhalational anesthesia is thought to modulate the immune system in a pro-cancerous way, while propofol may have opposite effects. Many of these recent studies are statistically underpowered and susceptible to bias, and experts in cancer treatment and anesthesia have emphasized the need for further research within this specific field.

In this study the investigators aim to characterize differences in the immunologic response to surgery between patients anesthetized with TIVA, epidural and NSAID and patients anesthetized with total intravenous anesthesia alone. This will be done by analyzing blood samples obtained in the perioperative period in patients undergoing different modes of anesthesia. The Investigators will furthermore describe the quality of recovery for patients anesthetized with the different methods Objectives The investigators hypothesize that the immunologic response to surgery and metastasis progression are influenced by the anesthetic technique.

Methods The study is initiated by Center for Surgical Science, Department of Surgery, Zealand University Hospital.

The study will take place at Hvidovre Hospital. This is a Danish university hospital. It supports 500,000 people and is one of four main emergency hospitals in Copenhagen Denmark. About 300 laparoscopic colon resections are performed at this facility every year.

Intervention Participants will undergo laparoscopic colon resection for cancer. They will be anaesthetized according to the standard operating procedure at Hvidovre Hospital with the exception that no dexamethasone is administered as it could modulate the immune response. This includes anesthesia induction and maintenance with intravenous propofol and remifentanil. Patients will receive 4 mg ondansetron at the end of anesthesia.

A thoracic epidural catheter will be installed preoperatively and kept for up to three days. After an initial bolus with bupivacaine, continuous infusion of bupivacaine and sufentanil will be used to maintain the epidural analgesic effect. Postoperatively the epidural will be paused or discontinued if it is displaced or if side effects occur. It will only be re-installed if there is still need of neuraxial analgesia.

Patients will follow a standard Enhanced Recovery After Surgery (ERAS) protocol used at the facility.

Blood samples will be obtained before surgery and at four time points postoperatively and patient files will be assessed for adverse events within 30 days from surgery.

Withdrawal criteria:

Patients can be withdrawn from the study for any of the following reasons:

* Failure to adhere to the anesthesia intervention described above- including failure to install effective continuous epidural anesthesia.
* Adverse events after surgery Any complication over grade 2 in Clavien-Dindo (26) classification Blood transfusion Deep vein thrombosis or pulmonary embolism Anastomotic leak Acute renal failure Infection (wound infection or systemic infection) during the observation period.
* After consultation patients can be withdrawn due to withdrawal of informed consent to participate in the study at the patients' own request at any time for any reason.

Population:

Study group: The "Hvidovre population":

The investigators will include patients undergoing laparoscopic hemicolectomy for cancer scheduled for anesthesia with total intravenous anesthesia combined with epidural anesthesia on Hvidovre Hospital according to the intervention described above.

Control group: The "Zealand University Hospital population" The immunological and oxidative stress in relation to abdominal surgery (IMOX) study is ongoing at Zealand University Hospital, Roskilde. It is a prospective explorative study cohort that consists of 60 patients undergoing laparoscopic colorectal cancer surgery. The aim of the study is to characterize the immunological and oxidative stress response to surgery. Outcomes similar to the primary and secondary outcomes of the ANIMOX-study are included in the IMOX-study. Patients are already included in the IMOX-study and blood samples are collected and kept in a bio bank.

The investigators will retrieve data on our main outcomes from the IMOX study in our analysis. Only electronic data will be used and no biologic material will be transferred from the IMOX project to ANIMOX. The population will be stratified according to anesthetic technique, which, according to the standard operating procedure, is either total intravenous anesthesia with propofol and remifentanil or volatile anesthesia with sevoflurane combined with a fast acting opioid (remifentanil or sufentanil). Patients anaesthetized with other techniques including epidural or other regional blocks will be excluded from the analysis.

Biological samples To characterize the immunological response to surgery the investigators obtain blood samples for analysis on postoperative day -1, 1, 2, 3 and 10 (or at the visit on day 10-14 where pathology results are given).

Handling of blood samples Blood samples will be drawn by a trained professional and analyzed immediately at the standard lab facilities at Hvidovre Hospital and destroyed immediately hereafter. The results will be accessible in Sundhedsplatformen.

ELIGIBILITY:
Inclusion Criteria:

1. Patients over 18 years
2. Patients diagnosed with colorectal cancer (UICC stadium I-III) and scheduled for laparoscopic hemicolectomy.
3. ASA class I-III (Classification of the American Society of Anesthesiology)
4. Patients scheduled for anesthesia with propofol, remifentanil and epidural anesthesia.
5. Signed informed consent

Exclusion Criteria:

1. Known immune-defects
2. Patients undergoing neoadjuvant chemo or radiotherapy
3. History of previous cancer
4. Patients in immunomodulatory treatment within last 6 months
5. Daily oral or intravenous steroid-use
6. Patients that have undergone major surgery within one month before planned colon resection.

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: We will include patients undergoing laparoscopic hemicolectomy for cancer scheduled for anesthesia with total intravenous anesthesia combined with epidural anesthesia on Hvidovre Hospital
Sampling Method: Non-Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2020-06-04 (Estimated); Primary Completion 2020-12-31 (Estimated); Study Completion 2020-12-31 (Estimated)

PRIMARY OUTCOMES:
Changes in neutrophil to lymphocyte ratio from preoperatively to day 1 postoperatively | From preoperatively to day 1 postoperatively
  Changes in neutrophil to lymphocyte ratio from day 0 to day 1. The ratio will be estimated using absolute numbers from differential counts pre and postoperatively. A high neutrophil to lymfocyte ratio is related to poor outcome after cancer surgery

SECONDARY OUTCOMES:
Changes in quality of recovery-15 score from preoperatively to day 1 postoperatively. | Difference from preoperatively to day 1 postoperatively
  The QoR-15 questionnaire results in a score of 0-150 where a high score reflects good recovery.

CONTACTS AND LOCATIONS:
Locations (1):
- Hvidovre University hospital, Hvidovre, Capital Region, Denmark

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Demicheli R, Fornili M, Ambrogi F, Higgins K, Boyd JA, Biganzoli E, Kelsey CR. Recurrence dynamics for non-small-cell lung cancer: effect of surgery on the development of metastases. J Thorac Oncol. 2012 Apr;7(4):723-30. doi: 10.1097/JTO.0b013e31824a9022. PMID 22425921
- [Background] Demicheli R, Biganzoli E, Boracchi P, Greco M, Retsky MW. Recurrence dynamics does not depend on the recurrence site. Breast Cancer Res. 2008;10(5):R83. doi: 10.1186/bcr2152. Epub 2008 Oct 9. PMID 18844974
- [Background] Ciechanowicz SJ, Ma D. Anaesthesia for oncological surgery - can it really influence cancer recurrence? Anaesthesia. 2016 Feb;71(2):127-31. doi: 10.1111/anae.13342. Epub 2015 Dec 16. No abstract available. PMID 26669960
- [Background] Freeman J, Connolly C, Buggy D. Mechanisms of Metastasis of Solid Organ Tumors in the Perioperative Period. Int Anesthesiol Clin. 2016 Fall;54(4):29-47. doi: 10.1097/AIA.0000000000000124. No abstract available. PMID 27648889
- [Background] Horowitz M, Neeman E, Sharon E, Ben-Eliyahu S. Exploiting the critical perioperative period to improve long-term cancer outcomes. Nat Rev Clin Oncol. 2015 Apr;12(4):213-26. doi: 10.1038/nrclinonc.2014.224. Epub 2015 Jan 20. PMID 25601442
- [Background] Yamaguchi K, Takagi Y, Aoki S, Futamura M, Saji S. Significant detection of circulating cancer cells in the blood by reverse transcriptase-polymerase chain reaction during colorectal cancer resection. Ann Surg. 2000 Jul;232(1):58-65. doi: 10.1097/00000658-200007000-00009. PMID 10862196
- [Background] Demicheli R, Retsky MW, Hrushesky WJ, Baum M, Gukas ID. The effects of surgery on tumor growth: a century of investigations. Ann Oncol. 2008 Nov;19(11):1821-8. doi: 10.1093/annonc/mdn386. Epub 2008 Jun 10. PMID 18550576
- [Background] Coffey JC, Wang JH, Smith MJ, Bouchier-Hayes D, Cotter TG, Redmond HP. Excisional surgery for cancer cure: therapy at a cost. Lancet Oncol. 2003 Dec;4(12):760-8. doi: 10.1016/s1470-2045(03)01282-8. PMID 14662433
- [Background] Duff S, Connolly C, Buggy DJ. Adrenergic, Inflammatory, and Immune Function in the Setting of Oncological Surgery: Their Effects on Cancer Progression and the Role of the Anesthetic Technique in their Modulation. Int Anesthesiol Clin. 2016 Fall;54(4):48-57. doi: 10.1097/AIA.0000000000000120. No abstract available. PMID 27648890
- [Background] Bartal I, Melamed R, Greenfeld K, Atzil S, Glasner A, Domankevich V, Naor R, Beilin B, Yardeni IZ, Ben-Eliyahu S. Immune perturbations in patients along the perioperative period: alterations in cell surface markers and leukocyte subtypes before and after surgery. Brain Behav Immun. 2010 Mar;24(3):376-86. doi: 10.1016/j.bbi.2009.02.010. Epub 2009 Feb 28. PMID 19254757
- [Background] Tai LH, de Souza CT, Belanger S, Ly L, Alkayyal AA, Zhang J, Rintoul JL, Ananth AA, Lam T, Breitbach CJ, Falls TJ, Kirn DH, Bell JC, Makrigiannis AP, Auer RA. Preventing postoperative metastatic disease by inhibiting surgery-induced dysfunction in natural killer cells. Cancer Res. 2013 Jan 1;73(1):97-107. doi: 10.1158/0008-5472.CAN-12-1993. Epub 2012 Oct 22. PMID 23090117
- [Background] Zimmitti G, Soliz J, Aloia TA, Gottumukkala V, Cata JP, Tzeng CW, Vauthey JN. Positive Impact of Epidural Analgesia on Oncologic Outcomes in Patients Undergoing Resection of Colorectal Liver Metastases. Ann Surg Oncol. 2016 Mar;23(3):1003-11. doi: 10.1245/s10434-015-4933-1. Epub 2015 Oct 28. PMID 26511261
- [Background] Hiller JG, Hacking MB, Link EK, Wessels KL, Riedel BJ. Perioperative epidural analgesia reduces cancer recurrence after gastro-oesophageal surgery. Acta Anaesthesiol Scand. 2014 Mar;58(3):281-90. doi: 10.1111/aas.12255. Epub 2014 Jan 2. PMID 24383612
- [Background] Gottschalk A, Ford JG, Regelin CC, You J, Mascha EJ, Sessler DI, Durieux ME, Nemergut EC. Association between epidural analgesia and cancer recurrence after colorectal cancer surgery. Anesthesiology. 2010 Jul;113(1):27-34. doi: 10.1097/ALN.0b013e3181de6d0d. PMID 20508494
- [Background] Exadaktylos AK, Buggy DJ, Moriarty DC, Mascha E, Sessler DI. Can anesthetic technique for primary breast cancer surgery affect recurrence or metastasis? Anesthesiology. 2006 Oct;105(4):660-4. doi: 10.1097/00000542-200610000-00008. PMID 17006061
- [Background] Piegeler T, Schlapfer M, Dull RO, Schwartz DE, Borgeat A, Minshall RD, Beck-Schimmer B. Clinically relevant concentrations of lidocaine and ropivacaine inhibit TNFalpha-induced invasion of lung adenocarcinoma cells in vitro by blocking the activation of Akt and focal adhesion kinase. Br J Anaesth. 2015 Nov;115(5):784-91. doi: 10.1093/bja/aev341. PMID 26475807
- [Background] Byrne K, Levins KJ, Buggy DJ. Can anesthetic-analgesic technique during primary cancer surgery affect recurrence or metastasis? Can J Anaesth. 2016 Feb;63(2):184-92. doi: 10.1007/s12630-015-0523-8. PMID 26497721
- [Background] Shi QY, Zhang SJ, Liu L, Chen QS, Yu LN, Zhang FJ, Yan M. Sevoflurane promotes the expansion of glioma stem cells through activation of hypoxia-inducible factors in vitro. Br J Anaesth. 2015 May;114(5):825-30. doi: 10.1093/bja/aeu402. Epub 2014 Dec 9. PMID 25492570
- [Background] Luo X, Zhao H, Hennah L, Ning J, Liu J, Tu H, Ma D. Impact of isoflurane on malignant capability of ovarian cancer in vitro. Br J Anaesth. 2015 May;114(5):831-9. doi: 10.1093/bja/aeu408. Epub 2014 Dec 13. PMID 25501719
- [Background] Xu YJ, Li SY, Cheng Q, Chen WK, Wang SL, Ren Y, Miao CH. Effects of anaesthesia on proliferation, invasion and apoptosis of LoVo colon cancer cells in vitro. Anaesthesia. 2016 Feb;71(2):147-54. doi: 10.1111/anae.13331. Epub 2015 Dec 16. PMID 26669824
- [Background] Stollings LM, Jia LJ, Tang P, Dou H, Lu B, Xu Y. Immune Modulation by Volatile Anesthetics. Anesthesiology. 2016 Aug;125(2):399-411. doi: 10.1097/ALN.0000000000001195. PMID 27286478
- [Background] Wigmore TJ, Mohammed K, Jhanji S. Long-term Survival for Patients Undergoing Volatile versus IV Anesthesia for Cancer Surgery: A Retrospective Analysis. Anesthesiology. 2016 Jan;124(1):69-79. doi: 10.1097/ALN.0000000000000936. PMID 26556730
- [Background] Buggy DJ, Borgeat A, Cata J, Doherty DG, Doornebal CW, Forget P, Gottumukkala V, Gottschalk A, Gupta A, Gupta K, Hales TG, Hemmings HC, Hollmann MW, Kurz A, Ma D, Parat MO, Sessler DI, Shorten G, Singleton P. Consensus statement from the BJA Workshop on Cancer and Anaesthesia. Br J Anaesth. 2015 Jan;114(1):2-3. doi: 10.1093/bja/aeu262. Epub 2014 Aug 7. No abstract available. PMID 25104229
- [Background] Piegeler T, Beck-Schimmer B. Anesthesia and colorectal cancer - The perioperative period as a window of opportunity? Eur J Surg Oncol. 2016 Sep;42(9):1286-95. doi: 10.1016/j.ejso.2016.05.004. Epub 2016 May 24. PMID 27265039

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2019-05-23): https://cdn.clinicaltrials.gov/large-docs/84/NCT03974984/Prot_SAP_000.pdf